CLINICAL TRIAL: NCT04844970
Title: A Randomized, Double-blind, and Placebo Controlled Multicenter Phase II Trial Evaluating Anamorelin in the Prevention of Cancer Induced-Weight Loss and Anorexia in Patients Receiving First-line Treatment of Advanced Pancreatic Cancer
Brief Title: Anamorelin Study for Advanced Pancreatic Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study closure was initiated by the financial sponsor and agreed upon by the site PI. The study is closing because of low enrollment and insufficient funds.
Sponsor: Lahey Clinic (Other)
Collaborators: Helsinn Healthcare SA (Industry); Quartesian LLC (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: LHMC 20193054
Record Dates: First submitted 2021-03-09; First posted 2021-04-14 (Actual); Results first posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Metastatic Pancreatic Cancer
Keywords: Phase II; Randomized; double-blind; placebo-controlled; Anamorelin HCI; Cachexia; Anorexia; Weight loss; FAACT A/CS
MeSH Terms: conditions — Pancreatic Neoplasms; Cachexia; Anorexia; Weight Loss | interventions — anamorelin

STUDY DESIGN:
Intervention Model Description: One group receives Anamorelin, and the other group receives placebo.
Who Masked: Participant, Investigator
Masking Description: double-blind. Neither the investigator nor the participant would know the assigned drug/placebo
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Anamorelin (Experimental): Patients randomized to anamorelin HCL will take it daily for 24 weeks starting 3-5 days prior to chemotherapy
  Interventions: Drug: Anamorelin Hydrochloride
- Placebo (Placebo Comparator): Patients randomized to placebo will take it daily for 24 weeks starting 3-5 days prior to chemotherapy
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Anamorelin Hydrochloride — Anamorelin HCl is an orally-active selective ghrelin receptor agonist which has shown anabolic and appetite-stimulating effects.
  Arms: Anamorelin
Drug: Placebo — Anamorelin placebo
  Arms: Placebo

SUMMARY:
Multicenter, double-blind, randomized, placebo-controlled study to evaluate the efficacy and safety of anamorelin HCl. Approximately 100 subjects with advanced PDAC and cachexia will be randomized 1:1 to anamorelin HCl 100 mg or placebo, taken orally once daily (QD) for a total of 25 weeks. Subjects will be instructed to take the study drug at least 1 hour before their first meal of the day

DETAILED DESCRIPTION:
Anorexia and cachexia are common clinical sequelae of uncontrolled, metastatic cancer. These effects can impair physical function, reduce quality of life, impair tolerability of anticancer therapy, and reduce survival. Anorexia and cachexia are especially challenging problems in patients diagnosed with metastatic pancreatic cancer. With an annual incidence approaching 50,000 patients in the U.S. alone, pancreatic cancer has an annual mortality of approximately 40,000 patients with most individuals succumbing to their disease within two years. Between 70-80% of patients with metastatic pancreatic cancer experience cancer cachexia, which has been associated with reduced survival, increased risk of disease progression, and impaired chemotherapy tolerance.

Anamorelin HCl is an orally-active selective ghrelin receptor agonist which has shown anabolic and appetite-stimulating effects. Several randomized, double-blind, clinical trials in cancer patients have shown that anamorelin HCL is safe, efficacious and increases lean body mass, bodyweight, and appetite. Investigators propose to test anamorelin HCL administered with chemotherapy in the first-line treatment of locally advanced unresectable and metastatic pancreatic cancer.

The study is a randomized, placebo controlled multicenter, Phase II trial to evaluate the efficacy and safety of anamorelin HCl. Approximately 100 patients with be enrolled in a 1:1 randomization to anamorelin HCL 100mg per day given concurrently with first-line chemotherapy compared to chemotherapy alone. Patients randomized to anamorelin HCL will take it daily for 24 weeks starting one day prior to chemotherapy. All patients will undergo an assessment by a certified nutritionist at or prior to their first cycle of chemotherapy. Both body weight and appetite will be measured at enrollment as well as at the initiation of chemotherapy. Patients will be stratified by degree of weight loss in the six months prior to enrollment, choice of first-line chemotherapy, and by baseline score of 5-item Anorexia Symptom Scale.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent
2. Female or male ≥18 years of age
3. Documented histologic or cytologic diagnosis of American Joint Committee on Cancer (AJCC) unresectable or metastatic pancreatic adenocarcinoma
4. Body mass index < 20 kg/m2 with involuntary weight loss or >5% within 6 months prior to screening
5. Ongoing problems with appetite/eating associated with the underlying cancer, as determined by having score of ≤ 17 points on the 5-item Anorexia Symptom Scale and ≤ 37 points on the 12-item FAACT A/CS
6. Subjects eligible to receive first line palliative chemotherapy
7. ECOG performance status 0 or 1 at screening
8. Acceptable hepatic function as defined by total bilirubin < 1.6 mg/dl unless associated with Gilbert syndrome, then total bilirubin < 2 x ULN. AST (SGOT) and ALT (SGPT) ≤ 2.5 x ULN or if hepatic metastases are present ≤ 5 x ULN
9. Appropriate treatment with pancreatic enzyme replacement prior to trial initiation
10. Female subjects shall be:

    1. of non-childbearing potential or
    2. of childbearing potential using reliable contraceptive measures and having a negative urine pregnancy test within 24 hours prior to first dose of investigational product.
11. The patient must be willing and able to comply with the protocol tests and procedures All inclusion criteria will be checked at screening visit (Visit 1).

Exclusion Criteria:

1. Patient with other forms of pancreatic cancer (e.g. neuroendocrine tumors)
2. Patient undergoing major surgery within 4 weeks of randomization or plans to undergo major surgery during study period.
3. Women who are pregnant or breastfeeding
4. Patient with alternative cause of cachexia as determined by the investigator including: a) severe COPD requiring O2, b) severe heart failure (NYHA Class III- IV), c) second malignancy
5. Reversible causes of reduced food intake as determined by the investigator including but not limited to: severe mucositis (>=NCI CTCAE grade 3), mechanical obstruction, severe nausea, vomiting, or diarrhea (>=NCI CTCAE grade 3)
6. Patient unable to swallow pills
7. Patient with history of bariatric surgery, gastrectomy, or malabsorption disorder (gastritis, esophagitis)
8. Patient with recent use of CYP3A4 inhibitors
9. Patient with current daily use of therapies that may increase the QRS interval durations
10. Patient currently taking medications/compounds intended to increase appetite or decrease weight loss (e.g. testosterone, megestrol acetate, cannabis products, methylphenidate, corticosteroids, olanzapine, mirtazapine (allowed if >4 weeks of use as therapy for depression)
11. Patient with current use of tube feeding or parenteral feeding
12. Patient with pleural effusion requiring thoracentesis, pericardial effusion requiring drainage, edema or evidence of ascites
13. Patient with uncontrolled or significant cardiovascular disease, including:

    1. History of myocardial infarction within the past 3 months
    2. A-V block of second or third degree (may be eligible if currently have a pacemaker)
    3. Unstable angina
    4. Congestive heart failure within the past 3 months, if defined as NYHA class III-IV
    5. Any history of clinically significant ventricular arrhythmias (such as ventricular tachycardia, ventricular fibrillation, Wolff-Parkinson-White (WPW) syndrome, or torsade de pointes)
    6. Uncontrolled hypertension (blood pressure >150 mm Hg systolic and >95 mm Hg diastolic)
    7. Heart rate < 50 beats per minute on pre-entry electrocardiogram and patient is symptomatic
14. Patient with uncontrolled diabetes mellitus or unmonitored diabetes mellitus
15. Patient with uncontrolled pain.
16. Any condition, including the presence of laboratory abnormalities, which in the Investigator's opinion, places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study
17. Enrollment in a previous study with anamorelin HCl
18. Enrollment in another clinical trial during the time of this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-11-07 (Actual); Study Completion 2023-11-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Keith Stuart, Principal Investigator — Lahey Hospital & Medical Center
Locations (1):
- Lahey Hospital & Medical Center, Burlington, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Anamorelin: Patients randomized to anamorelin HCL or placebo will take it daily for 24 weeks starting 3-5 days prior to chemotherapy.
  Anamorelin Hydrochloride: Anamorelin HCl is an orally-active selective ghrelin receptor agonist which has shown anabolic and appetite-stimulating effects.
- Placebo: Patients randomized to anamorelin HCL or placebo will take it daily for 24 weeks starting 3-5 days prior to chemotherapy.
Period: Overall Study
Arm/Group | Anamorelin | Placebo
Started | 2 | 2
Completed | 0 | 1
Not Completed | 2 | 1
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Anamorelin | Placebo | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 0 | 1
  >=65 years | 1 | 2 | 3
Age, Continuous [Mean (Full Range); unit: years] | 57.5 [46 to 69] | 75.5 [73 to 78] | 66.5 [46 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 2 | 2 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 2 | 4
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 1 | 2 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Percent Weight Change From Baseline to Week 25
Description: Does anamorelin HCl dosed at 100mg per day vs. placebo demonstrate superiority on body weight gain and improvement in anorexia symptoms in patients undergoing first-line chemotherapy for incurable pancreatic cancer.
Time Frame: 25 weeks from baseline
Population: No patients were analyzed for this outcome measure because no weight was collected at the 25-week time point.
Arm/Group | Anamorelin | Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Anorexia Questionnaire
Description: Absolute change in the Functional Assessment of Anorexia/Cachexia Treatment (FAACT 5) item Anorexia Symptom Score from baseline at week 13
Time Frame: from baseline to week 13
Population: Upon review of collected data, no subjects completed the FAACT - 5 questionnaire at the week 13 visit. Three out of 4 patient were not on the study at the week 13 visit.
Arm/Group | Anamorelin | Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Survival
Description: Overall Survival
Time Frame: 25 weeks
Population: Unable to analyze the Anamorelin group since both patients withdrew consent. One patient in the Placebo arm ended the study prior to week 13 and could not be analyzed for this outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Anamorelin | Placebo
Number analyzed (Participants) | 0 | 1
Participants |  | 1

4. Secondary Outcome: Radiologic Response to Chemotherapy
Description: Chemotherapy response will be evaluated by RECIST criteria
Time Frame: from baseline to week 13
Population: RECIST data was not collected for any patient at the week 13 time point and therefore not analyzed for this outcome. Three out of the 4 patients were not on the study at week 13, and one patient's RECIST data was not collected due to site error.
Arm/Group | Anamorelin | Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Weight Gain
Time Frame: from baseline to week 25 (end of the study)
Population: Weight was not collected for 3 out of 4 patients since they were already removed from the trial by week 25 and the fourth patients' weight was not collected due to site error.
Arm/Group | Anamorelin | Placebo
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Fatigue Questionnaire
Description: Change in Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F) questionnaire, fatigue subscale
Time Frame: from baseline to week 13
Population: Upon review of collected data, 3 of 4 patients were no longer on the trial at week 13. The fourth patients' data was not collected.
Arm/Group | Anamorelin | Placebo
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Number of Participants With Treatment-related Adverse Events as Assessed by CTCAE v5.0
Description: expected toxicities for Chemotherapies (FOLFIRINOX and Gemcitabine/Nab-Paclitaxel) will be assessed by CTCAE v5.0
Time Frame: from baseline to week 25 (end of study)
Population: 2 patients on the anamorelin arm both withdrew, data was collected until withdraw of consent. One patient on the placebo arm ended the study prior to week 13 (data collected up until they ended) and another patient's data was analyzed through week 25.
Measure: Count of Participants; unit: Participants
Arm/Group | Anamorelin | Placebo
Number analyzed (Participants) | 2 | 2
Participants | 0 | 1

8. Secondary Outcome: Adverse Events
Description: Number of AEs that are definitely related to Anamorelin or Placebo.
Time Frame: from baseline to week 25 (end of study)
Population: as for outcome 7
Measure: Number; unit: of events
Arm/Group | Anamorelin | Placebo
Number analyzed (Participants) | 2 | 2
of events | 0 | 0

9. Other Pre Specified Outcome: Unplanned Visits
Description: Number of unplanned visits for symptom management as defined by unscheduled clinic visits, emergency department visits, or hospitalizations
Time Frame: From baseline to week 25 (end of the study)
Population: Data for this outcome was not collected for any patient; no patients were analyzed.
Arm/Group | Anamorelin | Placebo
Number analyzed (Participants) | 0 | 0

10. Other Pre Specified Outcome: Chemotherapy Dose Change
Description: Percent change in dose intensity of chemotherapy as defined by percent reduction in anticipated chemotherapy dose as determined by the treating physician.
Time Frame: from baseline to week 13
Population: Chemotherapy dose change data was not collected for any patient. This outcome measure was not analyzed.
Groups:
- Anamorelin or Placebo: Patients randomized to anamorelin HCL or placebo will take it daily for 24 weeks starting 3-5 days prior to chemotherapy.
  Anamorelin Hydrochloride: Anamorelin HCl is an orally-active selective ghrelin receptor agonist which has shown anabolic and appetite-stimulating effects.
Arm/Group | Anamorelin or Placebo | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: AE data was to be collected from time of consent through the Week 25 visit. Patients on the anamorelin arm both withdrew, data was collected until withdraw of consent. One patient on the placebo arm ended the study prior to week 13 (data collected up until they ended) and another patients data was analyzed through week 25.
Description: AE definitions do not differ.
Arm/Group | Anamorelin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/2 | 1/2
Serious Adverse Events (participants affected / at risk) | 0/2 | 1/2
Other Adverse Events (participants affected / at risk) | 0/2 | 1/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anamorelin (N=2) | Placebo (N=2)
fatigue (General disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anamorelin (N=2) | Placebo (N=2)
confusion (Psychiatric disorders) | 0 (0) | 1 (1)
dizziness (Nervous system disorders) | 0 (0) | 1 (1)
hematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
ascities (Gastrointestinal disorders) | 0 (0) | 1 (1)
fatigue (General disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
This study closed to accrual early, with the limited number of participants, we were unable to analyze the data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-09-18): https://cdn.clinicaltrials.gov/large-docs/70/NCT04844970/Prot_SAP_000.pdf